CLINICAL TRIAL: NCT04306861
Title: Novel Multi-parametric MRI Techniques for Assessment of Patients With Pancreatic Ductal Adenocarcinoma Before and During Neoadjuvant Therapy
Brief Title: Novel MRI Techniques for Pancreatic Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Enrollment and other trial activities have temporarily paused due to COVID-19 and are expected to resume in the future; This is not a suspension of IRB approval
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Leo L Tsai, Assistant Professor of Radiology, Beth Israel Deaconess Medical Center
Other Study IDs: 2019-P-000549
Record Dates: First submitted 2019-11-22; First posted 2020-03-13 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Imaging; MRI; PDAC; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment Naïve PDAC Patients: Patient presenting with treatment-naïve, biopsy-proven pancreatic ductal adenocarcinoma (PDAC) who qualifies for neoadjuvant chemo-radiation therapy.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Baseline contrast-enhanced MRI and 2 follow-up contrast-enhanced MRIs (mid-treatment and treatment completion)

SUMMARY:
The purpose of this study is to optimize magnetic resonance imaging (MRI) sequences for imaging pancreatic ductal adenocarcinoma and correlate MRI biomarkers with the expression of the tumor suppressor gene SMAD4 and clinical outcomes with the goal of identifying which biomarkers are predictive of treatment response or non-response. This study will test magnetic resonance techniques on FDA approved clinical MRI machines in treatment-naïve patients with biopsy-proven PDAC.

DETAILED DESCRIPTION:
Specific Aims

1. To optimize the following multiparametric MRI sequences for imaging of Pancreatic ductal adenocarcinoma (PDAC): Arterial Spin Labeling (ASL), Blood Oxygenation Level Dependent (BOLD), Magnetization Transfer (MT), and reduced field-of-view Diffusion Weighted Imaging (DWI, including low b-values for intravoxel incoherent motion measurements and high b-values for Diffusion Kurtosis analysis).
2. To measure these MRI biomarkers in 20 treatment-naïve patients with biopsy-proven PDAC who have been referred to the Beth Israel Deaconess Medical Center (BIDMC) Pancreatic Cancer Program for neoadjuvant chemo-radiation therapy (CRT).
3. To correlate these MRI biomarkers with histopathology, i.e. the expression of the tumor suppressor gene SMAD4 and clinical outcomes with the goal of identifying which biomarkers are predictive of treatment response or non-response.

The investigators hypothesize the following:

1. It is feasible to develop dedicated MRI protocols with novel MRI techniques including Arterial Spin Labeling (ASL), Blood Oxygenation Level Dependent (BOLD), Magnetization Transfer (MT), and reduced field-of-view Diffusion Weighted Imaging (DWI), and to develop appropriate evaluation methods.
2. The implementation of these new protocols and evaluation methods in patients with pancreatic ductal adenocarcinoma (PDAC) provide biomarkers which correlate with histology and outcome in treatment-naïve patients.
3. The biomarkers are also predictive of therapy response in patients with PDAC during neoadjuvant chemo-radiation therapy (CRT) and correlate with the expression of the tumor suppressor gene SMAD4.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patient 18 years of age or older;
* Patient presenting with treatment-naïve, biopsy-proven pancreatic ductal adenocarcinoma (PDAC);
* Patient qualifying for neoadjuvant chemo-radiation therapy;
* Patient able and willing to participate in the study;
* Patient must sign the informed consent form in order to participate after the nature of the study has been fully explained to them and any questions they might have are adequately answered.
* eGFR levels greater than or equal to 30 mL/min/1.73m2 before contrast administration.

Exclusion Criteria:

* Patient previously-received or receiving treatment for PDAC at time of enrollment;
* Inability to understand or follow study instructions
* Diagnosed by a nutritionist with severe malnutrition;
* Unintentional weight loss of 20% or more throughout study;
* BMI of < 18.5;
* Patients with a contraindication to MRI examinations will be excluded from this study.
* Pregnancy
* Estimated Glomerular Filtration Rate (eGFR) levels < 30 mL/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient presenting with treatment-naïve, biopsy-proven pancreatic ductal adenocarcinoma (PDAC) who qualifies for neoadjuvant chemo-radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Optimize the following multiparametric MRI sequences for imaging of Pancreatic ductal adenocarcinoma (PDAC) | Study Duration, an average of 1 year
  Arterial Spin Labeling (ASL), Blood Oxygenation Level Dependent (BOLD), Magnetization Transfer (MT), and reduced field-of-view Diffusion Weighted Imaging (DWI, including low b-values for intravoxel incoherent motion measurements and high b-values for Diffusion Kurtosis analysis).
Measure the biomarkers obtained with MRI in treatment-naïve patients with biopsy-proven PDAC | Study Duration, an average of 1 year
  Biomarkers are obtained from the following imaging methods: Arterial Spin Labeling (ASL), Blood Oxygenation Level Dependent (BOLD), Magnetization Transfer (MT), and reduced field-of-view Diffusion Weighted Imaging (DWI, including low b-values for intravoxel incoherent motion measurements and high b-values for Diffusion Kurtosis analysis).
Correlate MRI biomarkers with histopathology (the expression of the tumor suppressor gene SMAD4 and clinical outcomes with the goal of identifying which biomarkers are predictive of treatment response or non-response). | Study Duration, an average of 1 year
  Biomarkers are obtained from the following imaging methods: Arterial Spin Labeling (ASL), Blood Oxygenation Level Dependent (BOLD), Magnetization Transfer (MT), and reduced field-of-view Diffusion Weighted Imaging (DWI, including low b-values for intravoxel incoherent motion measurements and high b-values for Diffusion Kurtosis analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Leo L Tsai, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Key Statistics for Pancreatic Cancer — http://www.cancer.org/cancer/pancreatic-cancer/about/key-statistics.html